CLINICAL TRIAL: NCT02337608
Title: Phase II, Randomized, Double-Blind, Placebo-Controlled, Proof of Concept Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of GLPG1205 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Efficacy and Safety of GLPG1205 in Subjects With Active Ulcerative Colitis
Acronym: ORIGIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1205-CL-211; 2014-001893-32 (EudraCT Number)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Ulcerative Colitis
Keywords: moderate to severe ulcerative colitis; GLPG1205
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GLPG1205

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLPG1205 100mg QD (Experimental): GLPG1205 100mg daily dosing in the morning
  Interventions: Drug: GLPG1205
- Placebo (Placebo Comparator): Placebo daily dosing in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1205 — GLPG1205 daily dosing in the morning for 12 weeks
  Arms: GLPG1205 100mg QD
Drug: Placebo — placebo daily dosing in the morning daily for 12 weeks
  Arms: Placebo

SUMMARY:
* Approximately 60 patients suffering from moderate to severe ulcerative colitis will be evaluated for improvement of disease activity (efficacy) when taking GLPG1205 or matching placebo once daily for 12 weeks in addition to their stable background treatment.
* During the course of the study, patients will also be examined for any side effects that may occur (safety and tolerability), and the amount of GLPG1205 present in the blood (Pharmacokinetics) as well as the effects of GLPG1205 on disease- and mechanism of action-related parameters (Pharmacodynamics) in blood, stool and colonic biopsies will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 75 years
* Documented history of UC
* Presence of active UC for a minimum period of 14 days prior to screening and spread beyond the rectum, Mayo score ≥ 6 with rectal bleeding score ≥ 1 and endoscopy score ≥ 2
* Absence of infectious colitis
* Tumor necrosis factor alpha (TNFα) inhibitor-naive subjects should have failed at least 1 prior conventional therapy
* Continuation of concurrent treatment with oral steroids (≤30 mg prednisolone eq/day), immunosuppressants and 5-aminosalicylates at stable dose is allowed
* Female subjects must have a negative blood pregnancy test, unless they are surgically sterile, had a hysterectomy, or have been postmenopausal for at least 1 year
* Subjects will have to use highly effective contraceptive methods

Exclusion Criteria:

* History of sensitivity to any component of the study drug, or a history of drug or other allergy
* Any concurrent illness, condition, disability, or clinically significant abnormality that, in the investigator's opinion, represents a safety risk for the subject's participation, may affect the interpretation of data, or may prevent the subject from safely completing the assessments
* History of significant psychological, neurologic, hepatic, renal, endocrine, cardiovascular, GI (other than UC), pulmonary, or metabolic disease
* History of active infections requiring intravenous antibiotics within the past 4 weeks prior to screening.
* History of malignancy within the past 5 years; presence or history of intestinal malignancy
* History of bowel surgery within 6 months prior to screening; history of colon resection with < 30 cm of the colon remaining
* Suspicion of Crohn's disease, indeterminate colitis, microscopic colitis, ischemic colitis, diverticular disease-associated colitis, or radiation-induced colitis
* Subject who has received non-permitted UC therapies within specified timeframes, depending on the medication, as stated in the protocol
* Subject who is pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in Mayo score at Week 8 | Screening and Week 8
  To evaluate the efficacy of GLPG1205 in terms of changes in Mayo score comparing results at Week 8 with baseline between GLPG1205 treated subjects and placebo subjects

SECONDARY OUTCOMES:
Changes in partial Mayo score | From Screening to Week 12
  To evaluate the efficacy of GLPG1205 in terms of changes in partial Mayo score comparing results with baseline between GLPG1205 treated subjects and placebo subjects at every visit up to Week 12
Histological response rate | Screening and Week 8
  To evaluate the efficacy of GLPG1205 in terms of histological response rate by use of the histopathological Geboes index comparing results at Week 8 with baseline between GLPG1205 treated subjects and placebo subjects
Number of subjects with adverse events | From Screening to Week 16
  To evaluate the safety and tolerability of GLPG1205 between GLPG1205 treated subjects and placebo subjects in terms of adverse events at every visit
Number of subjects with abnormal laboratory parameters | From Screening to Week 16
  To evaluate the safety and tolerability of GLPG1205 between GLPG1205 treated subjects and placebo subjects in terms of abnormal laboratory parameters at every visit
Number of subjects with abnormal vital signs | From Screening to Week 16
  To evaluate the safety and tolerability of GLPG1205 between GLPG1205 treated subjects and placebo subjects in terms of abnormal vital signs at every visit
Number of subjects with abnormal electrocardiogram | From Screening to Week 16
  To evaluate the safety and tolerability of GLPG1205 between GLPG1205 treated subjects and placebo subjects in terms of abnormal electrocardiograms at every visit
Number of subjects with abnormal physical examination | From Screening to Week 16
  To evaluate the safety and tolerability of GLPG1205 between GLPG1205 treated subjects and placebo subjects in terms of abnormal physical examination at every visit
The plasma levels of GLPG1205 | Week 4, 8 and 12
  To characterize the pharmacokinetics (PK) of GLPG1205 by measuring the amount in plasma at Week 4, 8 and 12
Changes in serum C-reactive protein (CRP) levels | From Screening to Week 16
  To characterize the pharmacodynamics (PD) of GLPG1205 by measuring the levels of C-reactive protein in serum at every visit
Changes in faecal calprotectin levels | From Screening to Week 12
  To characterize the pharmacodynamics (PD) of GLPG1205 by measuring the levels of faecal calprotectin in stool at every visit up to Week 12
Changes in myeloperoxidase (MPO) levels in colonic biopsies | Screening and Week 8
  To characterize the pharmacodynamics (PD) of GLPG1205 by measuring the levels of myeloperoxidase (MPO) in colonic biopsies at Screening and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (39):
- Belgium (3):
  - St. Pierre University Hospital Center, Brussels
  - Leuven University Hospital, Leuven
  - Clinic Saint-Joseph, Liège
- Czechia (5):
  - Hepato-Gastroenterology HK Ltd., Hradec Králové
  - Outpatient Clinic of Internal Medicine and Gastroenterology, Pilsen
  - Orlickoustecka Hospital, Inc., Ústí nad Orlicí
  - Regional Hospital T. Bata, Clinic of Internal Medicine, Zlín
  - Hospital Znojmo, Znojmo
- Germany (7):
  - Gastroenterology Specialist Practice, Berlin
  - Asklepios West Hospital Hamburg, Clinic of Internal Medicine, Hamburg
  - Hannover Medical School, Hanover
  - University Hospital Jena, Jena
  - Gastroenterology Group Practice Minden, Minden
  - Gastroenterology Practice at Germania-Campus, Münster
  - Internal Medicine Group Practice Oldenburg, Oldenburg
- Hungary (6):
  - Clinexpert Medical Center, Budapest
  - Hungarian Center for Obesity Ltd., Budapest
  - Medical Centre, Hungarian Defence Forces, Budapest
  - Szent Margit Hospital, Budapest
  - Main Railway Outpatient Clinic Debrecen, Debrecen
  - Javorszky Odon Hospital, Vác
- Poland (7):
  - Healthcare Center Orkan Med Stec Michalska Spolka Jawna, Ksawerów
  - Saint Family Hospital Medical Center, Lodz
  - Sopmed Llc, Sopot
  - H-T Medical Center, Tychy
  - Maternal, Pediatric and Adolescent Healtcare Centre, Gastroenterology Diagnostic Facility for Adults, Warsaw
  - Vivamed, Warsaw
  - Active Health Center, Non-Public Healthcare Facility Zawidawie Center, Wroclaw
- Russia (11):
  - Kazan State Medical University, Kazan'
  - Territorial Clinical Hospital, Krasnoyarsk
  - Central Research Institute of Gastroenterology, Moscow
  - Moscow Vladimirsky Regional Clinical Research Institute, Moscow
  - Semashko Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - City Clinical Hospital #12, Novosibirsk
  - Penza Regional Clinical Hospital n.a. N. N. Burdenko, Penza
  - City Clinical Hospital #31, Saint Petersburg
  - City General Hospital #2, Saint Petersburg
  - St. Venerable Martyress Elizabeth Municipal Hospital, Saint Petersburg
  - Stavropol State Medical University, Stavropol